CLINICAL TRIAL: NCT02931006
Title: Influence of Bovine Milk Consumption on Hormonal Profile in Males
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Bovine Milk-HMO-CTIL
Record Dates: First submitted 2016-09-15; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-09

CONDITIONS: Gonadotrophin and Sex Hormone Changes
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Placebo Comparator)
  Interventions: Other: water
- experimental (Active Comparator)
  Interventions: Other: bovine milk

INTERVENTIONS:
Other: water
  Arms: control
Other: bovine milk
  Arms: experimental

SUMMARY:
50 men will be recruited to this study. Participants will be asked to ingest commercially available bovine milk. Hormonal profile will be analyzed before and after consumption.

ELIGIBILITY:
Inclusion Criteria:

* healthy, non infertile males

Exclusion Criteria:

* lactose intolerance

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
sex hormone profile | 4 hours after consumption
  gonadotropin levels (Testosterone, Estradiol)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided